CLINICAL TRIAL: NCT05100381
Title: Effectiveness of Dry Needling on Pain, Functional Disability, Postural Control and Pain Pressure Threshold in Patients With Chronic Nonspecific Low Back Pain: A Double-Blind Randomised Controlled Trial
Brief Title: Effectiveness of Dry Needling in Patients With Chronic Nonspecific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1400.476
Record Dates: First submitted 2021-10-08; First posted 2021-10-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: dry needling; Low Back Pain; functional disability; postural control; pain pressure threshold
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will comprise 20 participants with chronic non-specific low back pain. The treatment will include dry needling of the lumbar multifidus muscle and routine physical therapy. The needles will be inserted to obtain local twitch response, and this process will continue until no more local twitch response occurs in each session. Then the needles will be left in place for 20 minutes. Routine physical therapy will include low level laser therapy and motor control training. The treatment will last 3 weeks, 6 sessions, twice a week.
  Interventions: Other: dry needling
- Control group (Placebo Comparator): The control group will comprise 20 participants with chronic non-specific low back pain. The treatment will include "sham" dry needling of the lumbar multifidus muscle and routine physical therapy. The sham dry needling method consists of the insertion of the needles subcutaneously and no local twitch response will be obtained. The needles will be left in the place for 20 minutes. Routine physical therapy will include low level laser therapy and motor control training. The treatment will last 3 weeks, 6 sessions, twice a week.
  Interventions: Other: sham (placebo) dry needling

INTERVENTIONS:
Other: dry needling — The patients will be placed in a prone position with a pillow under their belly to accommodate lumbar lordosis. Two lengths of sterile, disposable, 0.30 mm x 75 mm and 0.30 mm x 50 mm solid filament needle (Tony, China) will be used in this study. The length of the needle for each participant will be selected based on the size of the participant. The needles will be inserted into the lumbar multifidus muscle, 1.5 - 2 cm lateral to the spinous process of two or three painful segments, perpendicular to lamina (after piercing the skin, needles are directed inferomedially). The needles will be inserted to obtain local twitch response, and this process will continue until no more local twitch response occurs in each session. Then the needles will be left in place for 20 minutes.
  Arms: Experimental group
Other: sham (placebo) dry needling — The sham dry needling method includes the insertion of the needles subcutaneously and no local twitch response will be obtained. The needles will be left in the place for 20 minutes.
  Arms: Control group

SUMMARY:
Low back pain is a major health problem that affects psychosocial, economical, functional and physical aspects of the patients' life. The aim of this study will be to investigate the effectiveness of dry needling on pain, functional disability, postural control and pain pressure threshold in patients with chronic nonspecific low back pain using a randomized controlled trial design.

Patients with chronic nonspecific low back pain will be randomly divided into two groups: Experimental group (dry needling and routine physical therapy) and control group (sham dry needling and routine physical therapy). Primary outcomes will be pain intensity and functional disability. Postural control and pain pressure threshold will be considered as secondary outcomes.

DETAILED DESCRIPTION:
Low back pain is a major health problem that affects psychosocial, economical, functional and physical aspects of the patients' life. Since patients with chronic low back pain have impaired postural control and this impairment can cause chronicity and recurrence of low back pain, it is important to evaluate the effectiveness of interventions on postural control in patients with low back pain. Previous studies have shown the effectiveness of dry needling on pain, functional disability and pain sensitivity in patients with low back pain. The effectiveness of dry needling on postural control is not fully known.

The aim of this study will be to investigate the effectiveness of dry needling on pain, functional disability, postural control and pain pressure threshold in patients with chronic nonspecific low back pain.

This study will be a double-blind randomized controlled trial. Forty patients with chronic nonspecific low back pain will be randomly divided into two groups: Experimental group (dry needling and routine physical therapy) and control group (sham dry needling and routine physical therapy). Primary outcomes will be pain intensity and functional disability. Postural control and pain pressure threshold will be considered as secondary outcomes. Outcomes will be assessed before and one week after the intervention.

All of the participants will be identified and recruited by posters and word-of-mouth from the university and the surrounding local communities. Eligible participants will be explained about the purpose and the examination involved in this investigation, and all eligible participants will sign a written informed consent before entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 to 45 years.
* Moderate pain at rest (between 30 and 60 in NPRS).
* Patients with trigger points in the lumbar multifidus muscle.
* Patients have the ability to speak and read Persian.

Exclusion Criteria:

* Currently taking anticoagulant medications
* Specific low back pain (Neurogenic low back pain, Spinal stenosis, cauda equina syndrome, spondylolisthesis, and Presence of any signs or symptoms of non-musculoskeletal pathology e.g. cancer, infection and fracture in low back and lower extremities based on paraclinical findings)
* Prior surgery to the lumbosacral spine
* Inability to obtain prone lying
* Severe malalignments in the cervical, thoracic, lumbar or pelvic region and the lower limbs
* History of uncorrected vision impairment, vestibular, hearing or cognitive impairments
* Leg length discrepancy which disturbs balance
* Systemic diseases, such as diabetes, fibromyalgia, rheumatoid arthritis, degenerative diseases and other rheumatoid diseases
* Needle phobia
* Sacroiliac pain as identified with six clinical tests: compression, distraction, sacral thrust, thigh thrust, Gaenslen's and FABER's

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain level | before intervention (baseline) and one week after intervention
  The 0-100 Numeric Pain Rating Scale (NPRS) will be used to evaluate changing in level of pain from the baseline to one week after the intervention. Zero indicates no pain and 100 indicates maximum pain that the patient experiences. The NPRS has the responsiveness to measure the level of pain in people with low back pain.
Functional disability | before intervention (baseline) and one week after intervention
  The Persian version of The Oswestry Disability Index will be used to evaluate changing in functional disability from the baseline to one week after intervention. This questionnaire includes 10 activities of daily living and a total score of 100. A score below 25 indicates the lowest level of disability, 25 to 50 moderate disability, 50 to 75 severe disability, and 75 to 100 acute disability. The validity and the reliability of the Persian version of this questionnaire has been shown in the previous studies.

SECONDARY OUTCOMES:
Postural control | before intervention (baseline) and one week after intervention
  The force platform (Germany, Kistler, 9260AA6) will be used to evaluate postural control from the baseline to one week after intervention. Postural control will be evaluated in four different trials in double-leg stance position: 1-Eyes open on a firm surface. 2-Eyes closed on a firm surface. 3-Eyes open on a foam surface. 4-Eyes closed on a foam surface. The duration of each trial will be 90 s, three times repetition, with one minute rest interval between each trial. The postural control variables in this investigation will be COP excursion in the anteroposterior and mediolateral direction, COP amplitude standard deviation (dispersion) in the anteroposterior and mediolateral direction, COP velocity standard deviation in the anteroposterior and mediolateral direction, mean velocity of COP, COP total area of excursion, COP plane phase in the anteroposterior and mediolateral direction, and COP total plane phase.
Pain Pressure Threshold | before intervention (baseline) and one week after intervention
  The pressure algometer will be used to evaluate the Pain Pressure Threshold (PPT). The patients will be placed in a prone position with a pillow under their belly to accommodate lumbar lordosis and the algometer will be applied perpendicular to the muscle belly of the lumbar multifidus, approximately 1.5 cm lateral to the spinous process of the painful segments. The patients will be asked to signal verbally after perception of force change from pressure to pain. The PPT at each location will be taken three times and the mean of three repetitions will be used for statistical analysis. The validity and reliability of the pressure algometer has been shown in previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Pourahmadi, PhD, Study Director — Rehabilitation Research Center, Department of Physical Therapy, School of Rehabilitation Sciences, Iran University of Medical Sciences, Tehran, Iran
Locations (1):
- Physical therapy clinic at rehabilitation center of Iran university of medical sciences, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
The data sets of this study will be available on a reasonable request to the corresponding author.

REFERENCES:
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Mousavi SJ, Akbari ME, Mehdian H, Mobini B, Montazeri A, Akbarnia B, Parnianpour M. Low back pain in Iran: a growing need to adapt and implement evidence-based practice in developing countries. Spine (Phila Pa 1976). 2011 May 1;36(10):E638-46. doi: 10.1097/BRS.0b013e3181fa1da2. PMID 21270691
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Chiarotto A, Boers M, Deyo RA, Buchbinder R, Corbin TP, Costa LOP, Foster NE, Grotle M, Koes BW, Kovacs FM, Lin CC, Maher CG, Pearson AM, Peul WC, Schoene ML, Turk DC, van Tulder MW, Terwee CB, Ostelo RW. Core outcome measurement instruments for clinical trials in nonspecific low back pain. Pain. 2018 Mar;159(3):481-495. doi: 10.1097/j.pain.0000000000001117. PMID 29194127
- [Background] Rabey M, Beales D, Slater H, O'Sullivan P. Multidimensional pain profiles in four cases of chronic non-specific axial low back pain: An examination of the limitations of contemporary classification systems. Man Ther. 2015 Feb;20(1):138-47. doi: 10.1016/j.math.2014.07.015. Epub 2014 Aug 12. PMID 25153893
- [Background] Morrisette DC, Cholewicki J, Logan S, Seif G, McGowan S. A randomized clinical trial comparing extensible and inextensible lumbosacral orthoses and standard care alone in the management of lower back pain. Spine (Phila Pa 1976). 2014 Oct 1;39(21):1733-42. doi: 10.1097/BRS.0000000000000521. PMID 25054648
- [Background] Luomajoki H, Moseley GL. Tactile acuity and lumbopelvic motor control in patients with back pain and healthy controls. Br J Sports Med. 2011 Apr;45(5):437-40. doi: 10.1136/bjsm.2009.060731. Epub 2009 Jun 23. PMID 19553222
- [Background] Ruhe A, Fejer R, Walker B. Center of pressure excursion as a measure of balance performance in patients with non-specific low back pain compared to healthy controls: a systematic review of the literature. Eur Spine J. 2011 Mar;20(3):358-68. doi: 10.1007/s00586-010-1543-2. Epub 2010 Aug 19. PMID 20721676
- [Background] Hodges PW, Tucker K. Moving differently in pain: a new theory to explain the adaptation to pain. Pain. 2011 Mar;152(3 Suppl):S90-S98. doi: 10.1016/j.pain.2010.10.020. Epub 2010 Nov 18. No abstract available. PMID 21087823
- [Background] Schelldorfer S, Ernst MJ, Rast FM, Bauer CM, Meichtry A, Kool J. Low back pain and postural control, effects of task difficulty on centre of pressure and spinal kinematics. Gait Posture. 2015 Jan;41(1):112-8. doi: 10.1016/j.gaitpost.2014.09.004. Epub 2014 Sep 20. PMID 25270326
- [Background] Koch C, Hansel F. Non-specific Low Back Pain and Postural Control During Quiet Standing-A Systematic Review. Front Psychol. 2019 Mar 22;10:586. doi: 10.3389/fpsyg.2019.00586. eCollection 2019. PMID 30967811
- [Background] Berenshteyn Y, Gibson K, Hackett GC, Trem AB, Wilhelm M. Is standing balance altered in individuals with chronic low back pain? A systematic review. Disabil Rehabil. 2019 Jun;41(13):1514-1523. doi: 10.1080/09638288.2018.1433240. Epub 2018 Jan 30. PMID 29382241
- [Background] Brumagne S, Cordo P, Verschueren S. Proprioceptive weighting changes in persons with low back pain and elderly persons during upright standing. Neurosci Lett. 2004 Aug 5;366(1):63-6. doi: 10.1016/j.neulet.2004.05.013. PMID 15265591
- [Background] Crossman K, Mahon M, Watson PJ, Oldham JA, Cooper RG. Chronic low back pain-associated paraspinal muscle dysfunction is not the result of a constitutionally determined "adverse" fiber-type composition. Spine (Phila Pa 1976). 2004 Mar 15;29(6):628-34. doi: 10.1097/01.brs.0000115133.97216.ec. PMID 15014272
- [Background] MacDonald D, Moseley LG, Hodges PW. Why do some patients keep hurting their back? Evidence of ongoing back muscle dysfunction during remission from recurrent back pain. Pain. 2009 Apr;142(3):183-188. doi: 10.1016/j.pain.2008.12.002. Epub 2009 Jan 30. PMID 19186001
- [Background] Mannion AF, Weber BR, Dvorak J, Grob D, Muntener M. Fibre type characteristics of the lumbar paraspinal muscles in normal healthy subjects and in patients with low back pain. J Orthop Res. 1997 Nov;15(6):881-7. doi: 10.1002/jor.1100150614. PMID 9497814
- [Background] Larson DJ, Brown SHM. The effects of trunk extensor and abdominal muscle fatigue on postural control and trunk proprioception in young, healthy individuals. Hum Mov Sci. 2018 Feb;57:13-20. doi: 10.1016/j.humov.2017.10.019. Epub 2017 Nov 7. PMID 29121507
- [Background] Ghamkhar L, Kahlaee AH. The effect of trunk muscle fatigue on postural control of upright stance: A systematic review. Gait Posture. 2019 Jul;72:167-174. doi: 10.1016/j.gaitpost.2019.06.010. Epub 2019 Jun 11. PMID 31207565
- [Background] Yalfani A, Raeisi Z, Koumasian Z. Effects of eight-week water versus mat pilates on female patients with chronic nonspecific low back pain: Double-blind randomized clinical trial. J Bodyw Mov Ther. 2020 Oct;24(4):70-75. doi: 10.1016/j.jbmt.2020.06.002. Epub 2020 Jun 27. PMID 33218568
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Funk MF, Frisina-Deyo AJ. Dry needling for spine related disorders: a scoping review. Chiropr Man Therap. 2020 May 11;28(1):23. doi: 10.1186/s12998-020-00310-z. PMID 32393383
- [Background] Griswold D, Wilhelm M, Donaldson M, Learman K, Cleland J. The effectiveness of superficial versus deep dry needling or acupuncture for reducing pain and disability in individuals with spine-related painful conditions: a systematic review with meta-analysis. J Man Manip Ther. 2019 Jul;27(3):128-140. doi: 10.1080/10669817.2019.1589030. Epub 2019 Mar 19. PMID 30935320
- [Background] Hu HT, Gao H, Ma RJ, Zhao XF, Tian HF, Li L. Is dry needling effective for low back pain?: A systematic review and PRISMA-compliant meta-analysis. Medicine (Baltimore). 2018 Jun;97(26):e11225. doi: 10.1097/MD.0000000000011225. PMID 29952980
- [Background] Koppenhaver SL, Walker MJ, Rettig C, Davis J, Nelson C, Su J, Fernandez-de-Las-Penas C, Hebert JJ. The association between dry needling-induced twitch response and change in pain and muscle function in patients with low back pain: a quasi-experimental study. Physiotherapy. 2017 Jun;103(2):131-137. doi: 10.1016/j.physio.2016.05.002. Epub 2016 May 20. PMID 27623385
- [Background] Koppenhaver SL, Walker MJ, Su J, McGowen JM, Umlauf L, Harris KD, Ross MD. Changes in lumbar multifidus muscle function and nociceptive sensitivity in low back pain patient responders versus non-responders after dry needling treatment. Man Ther. 2015 Dec;20(6):769-76. doi: 10.1016/j.math.2015.03.003. Epub 2015 Mar 13. PMID 25801100
- [Background] Dar G, Hicks GE. The immediate effect of dry needling on multifidus muscles' function in healthy individuals. J Back Musculoskelet Rehabil. 2016 Apr 27;29(2):273-278. doi: 10.3233/BMR-150624. PMID 26406203
- [Background] Kiesel KB, Uhl TL, Underwood FB, Rodd DW, Nitz AJ. Measurement of lumbar multifidus muscle contraction with rehabilitative ultrasound imaging. Man Ther. 2007 May;12(2):161-6. doi: 10.1016/j.math.2006.06.011. Epub 2006 Sep 14. PMID 16973400
- [Background] Hodges PW. Pain and motor control: From the laboratory to rehabilitation. J Electromyogr Kinesiol. 2011 Apr;21(2):220-8. doi: 10.1016/j.jelekin.2011.01.002. PMID 21306915
- [Background] Emami F, Yoosefinejad AK, Razeghi M. Correlations between core muscle geometry, pain intensity, functional disability and postural balance in patients with nonspecific mechanical low back pain. Med Eng Phys. 2018 Oct;60:39-46. doi: 10.1016/j.medengphy.2018.07.006. Epub 2018 Aug 1. PMID 30077486
- [Background] Behennah J, Conway R, Fisher J, Osborne N, Steele J. The relationship between balance performance, lumbar extension strength, trunk extension endurance, and pain in participants with chronic low back pain, and those without. Clin Biomech (Bristol). 2018 Mar;53:22-30. doi: 10.1016/j.clinbiomech.2018.01.023. Epub 2018 Jan 31. PMID 29407352
- [Background] Loizidis T, Nikodelis T, Bakas E, Kollias I. The effects of dry needling on pain relief and functional balance in patients with sub-chronic low back pain. J Back Musculoskelet Rehabil. 2020;33(6):953-959. doi: 10.3233/BMR-181265. PMID 32310156
- [Background] Griswold D, Gargano F, Learman KE. A randomized clinical trial comparing non-thrust manipulation with segmental and distal dry needling on pain, disability, and rate of recovery for patients with non-specific low back pain. J Man Manip Ther. 2019 Jul;27(3):141-151. doi: 10.1080/10669817.2019.1574389. Epub 2019 Feb 9. PMID 30935327
- [Background] Tellez-Garcia M, de-la-Llave-Rincon AI, Salom-Moreno J, Palacios-Cena M, Ortega-Santiago R, Fernandez-de-Las-Penas C. Neuroscience education in addition to trigger point dry needling for the management of patients with mechanical chronic low back pain: A preliminary clinical trial. J Bodyw Mov Ther. 2015 Jul;19(3):464-72. doi: 10.1016/j.jbmt.2014.11.012. Epub 2014 Nov 22. PMID 26118519
- [Background] Nogueira JF, Carrasco AC, Pelegrinelli ARM, Guenka LC, Silva MF, Dela Bela LF, Dias JM, Moura FA, McVeigh JG, Cardoso JR. Posturography Comparison and Discriminant Analysis Between Individuals With and Without Chronic Low Back Pain. J Manipulative Physiol Ther. 2020 Jun;43(5):469-475. doi: 10.1016/j.jmpt.2019.01.002. Epub 2020 Jul 24. PMID 32718710
- [Background] Karimi Ghasem Abad S, Akhbari B, Salavati M, Talebian Moghaddam S, Saeedi A, Seydi M, Ahangari M, Negahban H. Reliability of postural control during double-leg standing in subjects with nonspecific chronic low back pain: Dual-task paradigm and manipulated visual and somatosensory inputs. J Bodyw Mov Ther. 2021 Apr;26:49-56. doi: 10.1016/j.jbmt.2020.09.005. Epub 2020 Sep 17. PMID 33992286
- [Background] da Silva RA, Vieira ER, Fernandes KBP, Andraus RA, Oliveira MR, Sturion LA, Calderon MG. People with chronic low back pain have poorer balance than controls in challenging tasks. Disabil Rehabil. 2018 Jun;40(11):1294-1300. doi: 10.1080/09638288.2017.1294627. Epub 2017 Mar 10. PMID 28282992
- [Background] Wang-Price S, Zafereo J, Couch Z, Brizzolara K, Heins T, Smith L. Short-term effects of two deep dry needling techniques on pressure pain thresholds and electromyographic amplitude of the lumbosacral multifidus in patients with low back pain - a randomized clinical trial. J Man Manip Ther. 2020 Dec;28(5):254-265. doi: 10.1080/10669817.2020.1714165. Epub 2020 Jan 17. PMID 31960773
- [Background] Liu L, Huang QM, Liu QG, Thitham N, Li LH, Ma YT, Zhao JM. Evidence for Dry Needling in the Management of Myofascial Trigger Points Associated With Low Back Pain: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Jan;99(1):144-152.e2. doi: 10.1016/j.apmr.2017.06.008. Epub 2017 Jul 8. PMID 28690077
- [Background] Gerwin RD, Shannon S, Hong CZ, Hubbard D, Gevirtz R. Interrater reliability in myofascial trigger point examination. Pain. 1997 Jan;69(1-2):65-73. doi: 10.1016/s0304-3959(96)03248-4. PMID 9060014
- [Background] Chou LW, Kao MJ, Lin JG. Probable mechanisms of needling therapies for myofascial pain control. Evid Based Complement Alternat Med. 2012;2012:705327. doi: 10.1155/2012/705327. Epub 2012 Dec 31. PMID 23346211
- [Background] Ylinen J. Pressure algometry. Aust J Physiother. 2007;53(3):207. doi: 10.1016/s0004-9514(07)70032-6. No abstract available. PMID 17899675
- [Background] Richter P, Werner J, Heerlein A, Kraus A, Sauer H. On the validity of the Beck Depression Inventory. A review. Psychopathology. 1998;31(3):160-8. doi: 10.1159/000066239. PMID 9636945
- [Background] Ghassemzadeh H, Mojtabai R, Karamghadiri N, Ebrahimkhani N. Psychometric properties of a Persian-language version of the Beck Depression Inventory--Second edition: BDI-II-PERSIAN. Depress Anxiety. 2005;21(4):185-92. doi: 10.1002/da.20070. PMID 16075452
- [Background] Vasheghani-Farahani A, Tahmasbi M, Asheri H, Ashraf H, Nedjat S, Kordi R. The Persian, last 7-day, long form of the International Physical Activity Questionnaire: translation and validation study. Asian J Sports Med. 2011 Jun;2(2):106-16. doi: 10.5812/asjsm.34781. PMID 22375226
- [Background] Pourahmadi MR, Bagheri R, Jannati E, Ebrahimi Takamjani I, Sarrafzadeh J, Mohsenifar H. Effect of Elastic Therapeutic Taping on Abdominal Muscle Endurance in Patients With Chronic Nonspecific Low Back Pain: A Randomized, Controlled, Single-Blind, Crossover Trial. J Manipulative Physiol Ther. 2018 Sep;41(7):609-620. doi: 10.1016/j.jmpt.2017.10.019. Epub 2018 Aug 8. PMID 30098819
- [Background] Gholami Borujeni B, Yalfani A. Reduction of postural sway in athletes with chronic low back pain through eight weeks of inspiratory muscle training: A randomized controlled trial. Clin Biomech (Bristol). 2019 Oct;69:215-220. doi: 10.1016/j.clinbiomech.2019.09.006. Epub 2019 Sep 10. PMID 31614295
- [Background] Koch C, Garcia-Augundez A, Gobel S, Hansel F. A case control study to investigate differences in motor control between individuals with and without non-specific low back pain during standing. PLoS One. 2020 Jul 6;15(7):e0234858. doi: 10.1371/journal.pone.0234858. eCollection 2020. PMID 32628670
- [Background] Azadinia F, Ebrahimi-Takamjani I, Kamyab M, Asgari M, Parnianpour M. Effects of lumbosacral orthosis on dynamical structure of center of pressure fluctuations in patients with non-specific chronic low back pain: A randomized controlled trial. J Bodyw Mov Ther. 2019 Oct;23(4):930-936. doi: 10.1016/j.jbmt.2019.01.014. Epub 2019 Jan 31. PMID 31733785
- [Background] Shahvarpour A, Preuss R, Lariviere C. The effect of extensible and non-extensible lumbar belts on trunk postural balance in subjects with low back pain and healthy controls. Gait Posture. 2019 Jul;72:211-216. doi: 10.1016/j.gaitpost.2019.06.013. Epub 2019 Jun 20. PMID 31255888
- [Background] Laslett M. Evidence-based diagnosis and treatment of the painful sacroiliac joint. J Man Manip Ther. 2008;16(3):142-52. doi: 10.1179/jmt.2008.16.3.142. PMID 19119403
- [Background] Mahmoudzadeh A, Rezaeian ZS, Karimi A, Dommerholt J. The effect of dry needling on the radiating pain in subjects with discogenic low-back pain: A randomized control trial. J Res Med Sci. 2016 Oct 18;21:86. doi: 10.4103/1735-1995.192502. eCollection 2016. PMID 28163732
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] Boyce D, Wempe H, Campbell C, Fuehne S, Zylstra E, Smith G, Wingard C, Jones R. ADVERSE EVENTS ASSOCIATED WITH THERAPEUTIC DRY NEEDLING. Int J Sports Phys Ther. 2020 Feb;15(1):103-113. PMID 32089962
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Mousavi SJ, Parnianpour M, Mehdian H, Montazeri A, Mobini B. The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E454-9. doi: 10.1097/01.brs.0000222141.61424.f7. PMID 16778675
- [Background] Ruhe A, Fejer R, Walker B. The test-retest reliability of centre of pressure measures in bipedal static task conditions--a systematic review of the literature. Gait Posture. 2010 Oct;32(4):436-45. doi: 10.1016/j.gaitpost.2010.09.012. Epub 2010 Oct 13. PMID 20947353
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Vallone F, Benedicenti S, Sorrenti E, Schiavetti I, Angiero F. Effect of diode laser in the treatment of patients with nonspecific chronic low back pain: a randomized controlled trial. Photomed Laser Surg. 2014 Sep;32(9):490-4. doi: 10.1089/pho.2014.3715. PMID 25141218
- [Background] Abdelbasset WK, Nambi G, Alsubaie SF, Abodonya AM, Saleh AK, Ataalla NN, Ibrahim AA, Tantawy SA, Kamel DM, Verma A, Moawd SA. A Randomized Comparative Study between High-Intensity and Low-Level Laser Therapy in the Treatment of Chronic Nonspecific Low Back Pain. Evid Based Complement Alternat Med. 2020 Oct 28;2020:1350281. doi: 10.1155/2020/1350281. eCollection 2020. PMID 33178306
- [Background] Narouei S, Barati AH, Akuzawa H, Talebian S, Ghiasi F, Akbari A, Alizadeh MH. Effects of core stabilization exercises on thickness and activity of trunk and hip muscles in subjects with nonspecific chronic low back pain. J Bodyw Mov Ther. 2020 Oct;24(4):138-146. doi: 10.1016/j.jbmt.2020.06.026. Epub 2020 Jul 30. PMID 33218502